CLINICAL TRIAL: NCT04029402
Title: Molecular Analysis of Diabetic Kidney Disease Biopsies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Ottawa (Other); University of British Columbia (Other); University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: 16-118
Record Dates: First submitted 2019-07-21; First posted 2019-07-23 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Diabetic Nephropathies; Kidney Disease, Chronic
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic | interventions — Sequence Analysis, RNA; Shadowing Technique, Histology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic kidney disease: Patients with archived biopsies with a pathologic diagnosis of diabetic kidney disease, interstitial fibrosis/tubular atrophy, or nephrosclerosis.
  Interventions: Other: RNA sequencing
- Healthy controls: Potential living donors with archived biopsies performed as part of their donor workup and with no diagnostic abnormalities
  Interventions: Other: RNA sequencing

INTERVENTIONS:
Other: RNA sequencing — Transcriptomic analysis of kidney biopsy tissue, and linking with slope of eGFR decline
  Other Names: Histology; Slope of eGFR decline

SUMMARY:
Despite decades of research, the pathogenesis of human diabetic kidney disease remains largely unclear. Our goal is to use archived human kidney biopsy tissue from patients with and with diabetic nephropathy to identify new molecules that drive and/or protect against disease progression. We will use RNA sequencing to identify transcriptomic changes that associate with histologic and functional outcomes.

DETAILED DESCRIPTION:
RESEARCH OBJECTIVES A. To identify differences in transcription profiles obtained from residual kidney tissue which was obtained for clinical purposes.

B. To identify differences in transcription profile between patients whose loss of kidney function progresses rapidly (eGFR decline ≥4ml/min/year) and in whom it progresses more slowly (eGFR decline <4ml/min/year).

C. To identify differences in transcription profile between predominantly glomerular and predominantly tubulointerstitial histopathological types .

D. To identify new pathogenetic pathways that may become targets for therapeutic intervention

METHODS The planned study centres on the use of archival biopsy material that is superfluous to what is or would be needed for clinical care (01/01/1995 to 31/05/2018 , n= approximately 400-500). Archived samples will be collected from St. Michael's Hospital and a number of collaborating centres, including but not limited to University of British Columbia, the University of Manitoba, and the University of Ottawa.

RNA will be extracted from the biopsy material using either the core that has been used for immunofluorescence microscopy and is stored at -80˚C, and/or the core that is formalin-fixed, embedded in paraffin wax and stored at room temperature. The RNA thereby extracted will be subjected to detailed interrogation by RNASeq to quantify the expression level of mRNAs (transcriptome) and compare differences, as indicated in the research objectives detailed above. The transcriptome will then be related to the clinical course (eGFR decline) and histopathological changes, in addition to examining potentially pathogenetically important and that are amenable to therapeutic intervention.

Histopathology will also be performed and classified according to established systems.

Clinical information that would be retrieved from patients' medical records are listed below.

Clinical data

1. Age
2. Gender
3. Ethnicity
4. Diabetes history
5. Diabetes type: 1, 2
6. Retinopathy history
7. Smoking history
8. Medications
9. Comorbidities
10. Past medical history
11. Primary nephrologist Laboratory data (prior to biopsy, at biopsy and post-biopsy)
12. Renal function measures and calculations. For example:

    i. Serum creatinine, eGFR ii. Change in creatinine and eGFR iii. Urinary albumin:creatinine values and ratio (ACR) iv. Urine protein:creatinine values and ratio (PCR) v. Urinary protein excretion rate (UPEx) vi. Changes in ACR, PCR, UPEx
13. Diabetes measures and calculations. Biopsy data
14. Biopsy related data

Each site will locally maintain a confidential Master Linking Log.

De-identified data will be entered into a secure REDCap database that is hosted by St. Michael's Hospital.

ELIGIBILITY:
Inclusion Criteria (diabetic kidney disease cases):

* history of type 1 or type 2 diabetes
* at least 1 archived native kidney biopsy that demonstrates either pure diabetic kidney disease or features of non-specific vascular disease, including glomerulosclerosis, non-inflammatory vascular disease,
* sufficient remaining archived kidney biopsy tissue for RNA sequencing (100 um thick tissue section) and histologic analysis (PAS and Masson Trichrome staining)

Exclusion Criteria (diabetic kidney disease cases):

* less than 3 eGFR values post-biopsy
* latest recorded eGFR values less than 6 months post-biopsy

Inclusion Criteria (healthy controls):

- at least 1 native kidney disease biopsy with no diagnostic abnormality

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 1. Cases: A group of patients with diabetic kidney disease
  2. Controls: A group of healthy control patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Interstitial fibrosis | Baseline biopsy
  Extent of interstitial fibrosis in kidney biopsy assessed using a semi-quantitative scale on light microscopy of biopsy sections
Glomerulosclerosis | Baseline biopsy
  Extent of glomerulosclerosis in kidney biopsy assessed using a semi-quantitative scale on light microscopy of biopsy sections
Renal function change | Baseline biopsy
  Slope of eGFR decline

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - University of Ottawa, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No